CLINICAL TRIAL: NCT03693183
Title: A Double-Masked, Randomized, Single-Center Study Evaluating the Effect of 0.30% Ketorolac/0.80% HPMC, 0.80% HPMC and Vehicle on Symptoms of Dry Eye After Exposure to the Controlled Adverse Environment (CAE)
Brief Title: Efficacy Study of Ketorolac and HPMC to Treat Dry Eye
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-004-02
Record Dates: First submitted 2015-11-11; First posted 2018-10-02 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ketorolac; Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ketorolac/HPMC (Experimental): Drug: Ketorolac/HPMC Ophthalmic Solution
  1 drop administered in each eye 4 times per day for 2 days
  Interventions: Drug: Ketorolac/HPMC
- HPMC (Active Comparator): Drug: 0.80% Hydroxypropyl Methylcellulose(HMPC) Ophthalmic Solution
  1 Drop administered in each eye 4 times per day for 2 days
  Interventions: Drug: HPMC
- Vehicle (Placebo Comparator): Drug: Vehicle Ophthalmic Solution
  1 drop administered in each eye 4 times a day for 2 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ketorolac/HPMC — 0.30% Ketorolac/0.80%HPMC Ophthalmic solution administered 4 times per day for 2 days
  Other Names: Ketorolac/Hydroxypropyl Methylcellulose
  Arms: Ketorolac/HPMC
Drug: HPMC — 0.80% Hydroxypropyl Methylcellulose solution 4 times per day for 2 days
  Other Names: Hydroxypropyl Methylcellulose
  Arms: HPMC
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether ketorolac and Hydroxypropyl Methylcellulose are effective in the treatment of Dry Eye.

DETAILED DESCRIPTION:
This is a double masked, randomized study with approximately 45 subjects randomized to one of the three treatment arms at a single site. There are 5 visits over the course of 16 days.

Visit 1: Day -7 Visit 2: Day 0 Visit 3: Day 2 Visit 4: Day 7 Visit 5: Day 9

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent;
2. Are 18 years of age or older;
3. Are able and willing to follow instructions, including participation in study assessments, and can be present for the required study visits for the duration of the study;
4. Have a corrected visual acuity LogMar +0.7 (ETDRS) or better in each eye;
5. Have a reported history of dry eye in each eye;
6. Have a history of use of or a desire to use an eye drop for dry eye symptoms within the past 6 months;
7. Have a central corneal sensitivity score greater than 55 mm in each eye at Visit 1;
8. Have an average diary reported score for ocular discomfort, burning, dryness, grittiness, or stinging of ≥ 1.5 during the one week run-in period between Visits 1 and 2;
9. Have a greater than or equal to 1 fluorescein staining score in any region in at least one eye prior to exposure to the CAE at Visit 1;
10. Report greater than or equal 3 in worst symptom for all diary entries between visits 2 and 3
11. If female and of childbearing potential. Are not pregnant, nursing, or planning a pregnancy. Women of childbearing potential are required to have a negative urine pregnancy test at the screening and exit visits and agree to use an acceptable method of contraception for the duration of the study.

Exclusion Criteria:

1. Have contraindications to the use of the study medication(s);
2. Have a known allergy or sensitivity to the study medication(s) or their components;
3. Have anterior blepharitis, which is deemed clinically significant and/or likely to interfere with study parameters in the opinion of the investigator;
4. Are diagnosed with an ongoing ocular infection (bacterial, viral, or fungal) or active ocular inflammation (e.g., follicular conjunctivitis);
5. Wear contact lenses within 1 week of Visit 1 or throughout the duration of the study;
6. Have previously had laser in situ keratomileusis (LASIK) surgery;
7. Are currently taking any topical ophthalmic prescriptions or over-the-counter (OTC) solutions, artificial tears, gels or scrubs and cannot discontinue these medications 2 hours prior to Visit 1 and for the duration of the trial;
8. Have used Restasis® within 30 days of Visit 1;
9. Have a systemic disease, or uncontrolled medical condition, that in the opinion of the investigator could interfere with study measurements or subject compliance;
10. Are currently taking (at Visit 1) any medication known to cause ocular drying that has not been used on a stable dosing regimen for 30 days prior to Visit 1;
11. Are currently pregnant, nursing, or planning a pregnancy;
12. (For women of childbearing potential) Are unwilling to submit a urine sample for a pregnancy test at Visit 1 and at exit visit;
13. Have received another experimental drug or device within 30 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06-15 (Actual); Study Completion 2009-06-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ketorolac and HPMC on ocular discomfort using the Ora Calibra® Ocular Discomfort scale. | Day 0 through Day 9
  Evaluate the symptoms of Ketorolac and HPMC on ocular discomfort in subjects with dry eye syndrome.

SECONDARY OUTCOMES:
Efficacy of Ketorolac and HPMC on fluorescein staining using the Ora Calibra® scale. | Day 0 through Day 9
  Evaluate fluorescein staining of Ketorolac and HPMC in subjects with dry eye syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: H. Jerome Crampton, MD, Principal Investigator — Ophthalmic Reserach Associates
Locations (1):
- Ophthalmic Reserach Associates, Andover, Massachusetts, United States